CLINICAL TRIAL: NCT01579084
Title: Safety and Tolerability of AGN-199201 in Patients With Erythema Associated With Rosacea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199201-001
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Rosacea; Erythema
MeSH Terms: conditions — Rosacea; Erythema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- AGN-199201 Formulation A and B (Experimental): AGN-199201 Formulation A applied to one side of the face and Formulation B applied to the other side of the face twice daily.
  Interventions: Drug: AGN-199201 Formulation A; Drug: AGN-199201 Formulation B
- AGN-199201 Formulation B and C (Experimental): AGN-199201 Formulation B applied to one side of the face and Formulation C applied to the other side of the face twice daily.
  Interventions: Drug: AGN-199201 Formulation B; Drug: AGN-199201 Formulation C
- AGN-199201 Formulation C and A (Experimental): AGN-199201 Formulation C applied to one side of the face and Formulation A applied to the other side of the face twice daily.
  Interventions: Drug: AGN-199201 Formulation A; Drug: AGN-199201 Formulation C
- AGN-199201 Formulation A and Vehicle (Other): AGN-199201 Formulation A applied to one side of the face and AGN-199201 Vehicle applied to the other side of the face twice daily.
  Interventions: Drug: AGN-199201 Formulation A; Drug: AGN-199201 Vehicle
- AGN-199201 Formulation B and Vehicle (Other): AGN-199201 Formulation B applied to one side of the face and AGN-199201 Vehicle applied to the other side of the face twice daily.
  Interventions: Drug: AGN-199201 Formulation B; Drug: AGN-199201 Vehicle
- AGN-199201 Formulation C and Vehicle (Other): AGN-199201 Formulation C applied to one side of the face and AGN-199201 Vehicle applied to the other side of the face twice daily.
  Interventions: Drug: AGN-199201 Formulation C; Drug: AGN-199201 Vehicle
- AGN-199201 Formulation A (Experimental): AGN-199201 Formulation A applied to both sides of the face twice daily.
  Interventions: Drug: AGN-199201 Formulation A
- AGN-199201 Formulation B (Experimental): AGN-199201 Formulation B applied to both sides of the face twice daily.
  Interventions: Drug: AGN-199201 Formulation B
- AGN-199201 Formulation C (Experimental): AGN-199201 Formulation C applied to both sides of the face twice daily.
  Interventions: Drug: AGN-199201 Formulation C
- AGN-199201 Vehicle (Placebo Comparator): AGN-199201 Vehicle (Placebo) applied to both sides of the face twice daily.
  Interventions: Drug: AGN-199201 Vehicle

INTERVENTIONS:
Drug: AGN-199201 Formulation A — AGN-199201 Formulation A applied to the face as per protocol twice daily.
  Arms: AGN-199201 Formulation A; AGN-199201 Formulation A and B; AGN-199201 Formulation A and Vehicle; AGN-199201 Formulation C and A
Drug: AGN-199201 Formulation B — AGN-199201 Formulation B applied to the face as per protocol twice daily.
  Arms: AGN-199201 Formulation A and B; AGN-199201 Formulation B; AGN-199201 Formulation B and C; AGN-199201 Formulation B and Vehicle
Drug: AGN-199201 Formulation C — AGN-199201 Formulation C applied to the face as per protocol twice daily.
  Arms: AGN-199201 Formulation B and C; AGN-199201 Formulation C; AGN-199201 Formulation C and A; AGN-199201 Formulation C and Vehicle
Drug: AGN-199201 Vehicle — AGN-199201 vehicle (placebo) applied to the face as per protocol twice daily.
  Arms: AGN-199201 Formulation A and Vehicle; AGN-199201 Formulation B and Vehicle; AGN-199201 Formulation C and Vehicle; AGN-199201 Vehicle

SUMMARY:
This study will evaluate the safety and tolerability of AGN-199201 for the treatment of erythema associated with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* facial erythema associated with rosacea on both sides of the face

Exclusion Criteria:

* Laser light-source or other energy based therapy in the last 6 months
* Excessive hair around the treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AGN-199201 Formulation A and B: AGN-199201 Formulation A applied to one side of the face and Formulation B applied to the other side of the face twice daily for 5 days.
- AGN-199201 Formulation B and C: AGN-199201 Formulation B applied to one side of the face and Formulation C applied to the other side of the face twice daily for 5 days.
- AGN-199201 Formulation C and A: AGN-199201 Formulation C applied to one side of the face and Formulation A applied to the other side of the face twice daily for 5 days.
- AGN-199201 Formulation A and Vehicle: AGN-199201 Formulation A applied to one side of the face and AGN-199201 Vehicle applied to the other side of the face twice daily for 5 days.
- AGN-199201 Formulation B and Vehicle: AGN-199201 Formulation B applied to one side of the face and AGN-199201 Vehicle applied to the other side of the face twice daily for 5 days.
- AGN-199201 Formulation C and Vehicle: AGN-199201 Formulation C applied to one side of the face and AGN-199201 Vehicle applied to the other side of the face twice daily for 5 days.
- AGN-199201 Formulation A: AGN-199201 Formulation A applied to both sides of the face twice daily for 5 days.
- AGN-199201 Formulation B: AGN-199201 Formulation B applied to both sides of the face twice daily for 5 days.
- AGN-199201 Formulation C: AGN-199201 Formulation C applied to both sides of the face twice daily for 5 days.
- AGN-199201 Vehicle: AGN-199201 Vehicle (Placebo) applied to both sides of the face twice daily for 5 days.
Period: Overall Study
Arm/Group | AGN-199201 Formulation A and B | AGN-199201 Formulation B and C | AGN-199201 Formulation C and A | AGN-199201 Formulation A and Vehicle | AGN-199201 Formulation B and Vehicle | AGN-199201 Formulation C and Vehicle | AGN-199201 Formulation A | AGN-199201 Formulation B | AGN-199201 Formulation C | AGN-199201 Vehicle
Started | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 4
Completed | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-199201 Formulation A and B | AGN-199201 Formulation B and C | AGN-199201 Formulation C and A | AGN-199201 Formulation A and Vehicle | AGN-199201 Formulation B and Vehicle | AGN-199201 Formulation C and Vehicle | AGN-199201 Formulation A | AGN-199201 Formulation B | AGN-199201 Formulation C | AGN-199201 Vehicle | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 4 | 64
Age, Customized [Number; unit: Participants]
  < 45 years | 1 | 1 | 1 | 4 | 0 | 1 | 0 | 1 | 1 | 0 | 10
  45 to 65 years | 7 | 6 | 6 | 4 | 8 | 7 | 3 | 3 | 2 | 4 | 50
  > 65 years | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 6 | 7 | 5 | 7 | 2 | 4 | 2 | 3 | 49
  Male | 3 | 0 | 2 | 1 | 3 | 1 | 2 | 0 | 2 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders With at Least a 2-Grade Decrease From Baseline in Both Clinician Erythema Assessment (CEA) and Subject's Self Assessment (SSA) at Day 1
Description: The percentage of responders was determined by facial sides with at least a 2-grade decrease from Baseline (Improvement) in the CEA score and at least a 2-grade decrease from Baseline (Improvement) in the SSA score at Day 1. The investigator evaluated the severity of the participant's erythema (redness of the skin) as measured by the CEA using a 5-point scale where 0=clear skin with no signs of erythema; 1=almost clear of erythema, slight redness; 2=mild erythema, definite redness; 3=moderate erythema, marked redness and 4=severe erythema, fiery redness. The participant assessed the severity of their erythema as measured by the SSA using a 5-point scale where 0=clear of unwanted redness; 1=nearly clear of unwanted redness; 2=somewhat more redness than I prefer; 3=more redness than I prefer and 4=completely unacceptable redness.
Time Frame: Baseline, Day 1-hour 6
Population: Modified Intent-to-treat population consisted of all randomized patients who received study medication and who had measurements at Baseline and at least 1 post-baseline measurement for both CEA and SSA.
Measure: Number; unit: Percentage of responders
Units Other Than Participants: Facial Sides
Groups:
- AGN-199201 Formulation A: AGN-199201 Formulation A applied to the face twice daily for 5 days. Includes participants treated with Formulation A in any of the randomized treatment groups.
- AGN-199201 Formulation B: AGN-199201 Formulation B applied to the face twice daily for 5 days. Includes participants treated with Formulation B in any of the randomized treatment groups.
- AGN-199201 Formulation C: AGN-199201 Formulation C applied to the face twice daily for 5 days. Includes participants treated with Formulation C in any of the randomized treatment groups.
- AGN-199201 Vehicle: AGN-199201 Vehicle (Placebo) applied to the face twice daily for 5 days. Includes participants treated with Vehicle in any of the randomized treatment groups.
Arm/Group | AGN-199201 Formulation A | AGN-199201 Formulation B | AGN-199201 Formulation C | AGN-199201 Vehicle
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Facial Sides) | 32 | 32 | 32 | 32
Percentage of responders | 15.6 | 21.9 | 28.1 | 0.0

2. Secondary Outcome: Percentage of Responders With at Least a 2-Grade Decrease From Baseline on CEA
Description: The percentage of responders was determined by facial sides with at least a 2-grade decrease from Baseline (Improvement) in the CEA score at Day 1 and Day 5. The investigator evaluated the severity of the participant's erythema (redness of the skin) as measured by the CEA using a 5-point scale where 0=clear skin with no signs of erythema; 1=almost clear of erythema, slight redness; 2=mild erythema, definite redness; 3=moderate erythema, marked redness and 4=severe erythema, fiery redness.
Time Frame: Baseline, Day 1-hour 6, Day 5-hour 6
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Units Other Than Participants: Facial sides
Arm/Group | AGN-199201 Formulation A | AGN-199201 Formulation B | AGN-199201 Formulation C | AGN-199201 Vehicle
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Facial sides) | 32 | 32 | 32 | 32
Percentage of responders
  Day 1-hour 6 | 34.4 | 34.4 | 40.6 | 0.0
  Day 5-hour 6 (Facial Sides n=32,31,31,32) | 15.6 | 6.5 | 6.5 | 6.3

3. Secondary Outcome: Percentage of Responders With at Least a 2-Grade Decrease From Baseline on SSA
Description: The percentage of responders was determined by facial sides with at least a 2-grade decrease from Baseline (Improvement) in the SSA score at Day 1 and Day 5. The participant assessed the severity of their erythema as measured by the SSA using a 5-point scale where 0=clear of unwanted redness; 1=nearly clear of unwanted redness; 2=somewhat more redness than I prefer; 3=more redness than I prefer and 4=completely unacceptable redness.
Time Frame: Baseline, Day1-hour 6, Day 5-hour 6
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Units Other Than Participants: Facial sides
Arm/Group | AGN-199201 Formulation A | AGN-199201 Formulation B | AGN-199201 Formulation C | AGN-199201 Vehicle
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Facial sides) | 32 | 32 | 32 | 32
Percentage of responders
  Day1-hour 6 | 31.3 | 46.9 | 56.3 | 3.1
  Day 5-hour 6 (Facial Sides n=32,31,31,32) | 34.4 | 41.9 | 58.1 | 28.1

4. Primary Outcome: Percentage of Responders With at Least a 2-Grade Decrease From Baseline on Both Clinician Erythema Assessment (CEA) and Subject's Self Assessment (SSA) at Day 5
Description: The percentage of responders was determined by facial sides with at least a 2-grade decrease from Baseline (Improvement) in the CEA score and at least a 2-grade decrease from Baseline (Improvement) in the SSA score at Day 5. The investigator evaluated the severity of the participant's erythema (redness of the skin) as measured by the CEA using a 5-point scale where 0=clear skin with no signs of erythema; 1=almost clear of erythema, slight redness; 2=mild erythema, definite redness; 3=moderate erythema, marked redness and 4=severe erythema, fiery redness. The participant assessed the severity of their erythema as measured by the SSA using a 5-point scale where 0=clear of unwanted redness; 1=nearly clear of unwanted redness; 2=somewhat more redness than I prefer; 3=more redness than I prefer and 4=completely unacceptable redness.
Time Frame: Baseline, Day 5-hour 6
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Units Other Than Participants: Facial sides
Arm/Group | AGN-199201 Formulation A | AGN-199201 Formulation B | AGN-199201 Formulation C | AGN-199201 Vehicle
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Facial sides) | 32 | 31 | 31 | 32
Percentage of responders | 6.3 | 6.5 | 6.5 | 3.1

ADVERSE EVENTS:
Description: Serious Adverse Events and Adverse Events are reported by treatment arm not necessarily by individual intervention (treatment) received.
Arm/Group | AGN-199201 Formulation A and B | AGN-199201 Formulation B and C | AGN-199201 Formulation C and A | AGN-199201 Formulation A and Vehicle | AGN-199201 Formulation B and Vehicle | AGN-199201 Formulation C and Vehicle | AGN-199201 Formulation A | AGN-199201 Formulation B | AGN-199201 Formulation C | AGN-199201 Vehicle
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/8 | 5/8 | 3/8 | 6/8 | 6/8 | 4/8 | 3/4 | 3/4 | 3/4 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-199201 Formulation A and B (N=8) | AGN-199201 Formulation B and C (N=8) | AGN-199201 Formulation C and A (N=8) | AGN-199201 Formulation A and Vehicle (N=8) | AGN-199201 Formulation B and Vehicle (N=8) | AGN-199201 Formulation C and Vehicle (N=8) | AGN-199201 Formulation A (N=4) | AGN-199201 Formulation B (N=4) | AGN-199201 Formulation C (N=4) | AGN-199201 Vehicle (N=4)
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site anaesthesia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site dryness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site erosion (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Application site exfoliation (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Application site nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Application site pain (General disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0
Application site papules (General disorders) | 1 | 3 | 0 | 2 | 2 | 0 | 2 | 1 | 2 | 0
Application site paraesthesia (General disorders) | 1 | 2 | 2 | 2 | 0 | 1 | 0 | 2 | 0 | 0
Application site pruritus (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site warmth (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site pustules (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected bites (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 3 | 3 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.